CLINICAL TRIAL: NCT04936802
Title: Safety and Feasibility of the Transcatheter Tricuspid Valve Repair System (Trialign) for the Treatment or Reduction of Moderate to Severe Functional Tricuspid Regurgitation
Brief Title: Safety and Feasibility of the Transcatheter Tricuspid Valve Repair System (Trialign)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trialign study
Record Dates: First submitted 2021-06-03; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Tricuspid valve repair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcatheter tricuspid valve repair system (Trialign) (Experimental): Subjects who received transcatheter tricuspid valve repair with Trialign will be included in this arm.
  Interventions: Device: Transcatheter tricuspid valve repair system (Trialign)

INTERVENTIONS:
Device: Transcatheter tricuspid valve repair system (Trialign) — To assess the Trialign System to treat subjects with moderate to severe tricuspid regurgitation

SUMMARY:
The purpose of the study is to demonstrate safety and feasibility of the transcatheter tricuspid valve repair system (Trialign) for the treatment or reduction of moderate to severe functional tricuspid regurgitation.

DETAILED DESCRIPTION:
This study is a prospective single-arm trial for transcatheter tricuspid valve repair system (Trialign). A series of physical, imaging and laboratory exams will be performed to determine whether a subject has moderate to severe tricuspid regurgitation with high surgical risk. Subjects who meet the criteria will then receiveTrialign treatment if an informed consent is obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects has been informed the study and provided written informed consent.
2. Age ≥ 18 and ≤ 85 years old.
3. NYHA class II, III or ambulatory IV.
4. The subject was diagnosed moderate to severe functional tricuspid regurgitation
5. The subject was at high risk for open heart valve surgery. The heart team recommended tricuspid annuloplasty.
6. Subjects shall meet all selected criteria for TEE with moderate or severe tricuspid regurgitation.

   1. Systolic pulmonary artery pressure (SPAP) ≤ 60mmHg.
   2. Left ventricular ejection fraction (LVEF) ≥ 30%.
   3. Right ventricle tricuspid annular plane systolic excursion (TAPSE) ≥ 15 mm.
   4. Tricuspid valve annular diameter ≤ 55 mm.
   5. Tricuspid EROA ≤ 1.75 cm2.
   6. Functional tricuspid valve regurgitation pathology with a structurally normal valve.
7. Sufficient posterior annular dimension for device implantation.

Exclusion Criteria:

1. Severe uncontrolled hypertension (SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg).
2. History of heart transplant.
3. Previous tricuspid valve repair or replacement (including artificial valve).
4. Presence of a left ventricular assist device.
5. Active endocarditis.
6. Severe degenerative tricuspid valve disease.
7. Severe aortic stenosis.
8. The degree of mitral regurgitation is greater than grade 3.
9. Complete occlusion due to chronic calcification of the right coronary artery.
10. History of right internal jugular vein occlusion or thrombosis;
11. Anatomy in the region of the access path (right internal jugular vein) prevented correct placement of a percutaneous tricuspid valve annuloplasty system (e.g.: the presence of spinal stenosis, stent, vascular prosthesis).
12. An indication of the presence of thrombi in the right ventricle or atrium.
13. Myocardial infarction (MI) or known unstable angina within the 30 days prior to the index procedure.
14. Any percutaneous coronary intervention (PCI) within 30 days prior to the index procedure or planned 3 months post-the index procedure.
15. Hemodynamic instability or cardiogenic shock.
16. Restrictive or hypertrophic cardiomyopathy. Constructive pericarditis, or other structural heart disease.
17. Cerebrovascular accident (CVA) within the past 6 months
18. Serum creatinine > 2.5 mg/dL (or 221 μmol/L), Impaired kidney function, defined as glomerular filtration rate (GFR) of 30 mL/min or less.
19. Anemia (hemoglobin <<90g/L) not corrected by transfusion. Thrombocytopenia (platelet count <100×109/L) or thrombocytosis (>750×109/L).
20. Bleeding disorders or hypercoagulable state.
21. Active peptic ulcer or active gastrointestinal bleeding.
22. Contraindication to anticoagulant or antiplatelet therapies.
23. Contraindications to or refusal of blood transfusions.
24. Known allergy to stainless steel, nickel, platinum iridium, polyester and/or silk.
25. Pregnant or lactating; or female of childbearing potential with a positive pregnancy test 24 hours before any study-related radiation exposure.
26. Life expectancy less than 12 months.
27. Concurrent use of another clinical study product or use of another clinical study product within 30 days prior to enrolment.
28. Other circumstances deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-06-25 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Severe adverse device events (SADE) | 30 days
  Severe adverse device events (SADE) , defined as any device related complication, including but not limited to: death, myocardial infarction, stroke, reoperation, renal failure, pulmonary embolism, gastrointestinal bleeding, readmission, etc.

SECONDARY OUTCOMES:
Technical success | 30 days
  Technical success, defined as freedom from death with:
  1. Successful access, delivery and retrieval of the device delivery system;
  2. Deployment and correct positioning of the intended device(s) which is maintained and;
  3. No need for additional unplanned or emergency surgery or re-intervention related to the device or access procedure.
Evaluation of tricuspid valve function | 6 months
New York Heart Association (NYHA) classification | 6 months
6-minute walk test (6MWT) | 6 months
EuroQol five dimensions questionnaire (EQ-5D) | 6 months
Incidence of adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, Principal Investigator — Xijing Hospital

IPD SHARING:
Plan to Share IPD: No